CLINICAL TRIAL: NCT06495944
Title: An Open-Label, Single-Sequence Crossover, Drug-Drug Interaction Study to Characterize the Impact of the Cytochrome P450 3A Inhibitor Itraconazole on the Pharmacokinetics and Safety of Dazucorilant in Healthy, Adult Subjects
Brief Title: Impact of Itraconazole on the Pharmacokinetics and Safety of Dazucorilant in Healthy, Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CORT113176-655
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Healthy Adults
MeSH Terms: interventions — CORT113176; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dazucorilant (300 mg) and itraconazole (200 mg) (Experimental): On Days 1 and 8, each participant will receive a single oral dose of dazucorilant 300 mg, in a fed state. On Days 5-11, all participants will be administered once daily, oral doses of itraconazole 200 mg, in a fed state.
  Interventions: Drug: Dazucorilant; Drug: Itraconazole

INTERVENTIONS:
Drug: Dazucorilant — 75 mg soft gelatin capsules formulation for oral administration
  Other Names: CORT113176
Drug: Itraconazole — 100 mg capsules for oral administration

SUMMARY:
This study aims to answer how repeat doses of itraconazole impact the pharmacokinetics, safety, and tolerability of single doses of dazucorilant in healthy adults.

Participants in this study will complete screening assessments within 28 days before the first dose of study drug. Those participants who can participate will be admitted to the clinical pharmacology center (CPC) and complete pretreatment tests. Those participants will stay at the CPC for the duration of the study. On Days 1 and 8, each participant will receive a single oral dose of dazucorilant 300 mg, after eating. On Days 5-11, all participants will receive once daily, oral doses of itraconazole 200 mg, after eating. Blood and safety assessments will continue for 96-hours after dosing on Day 1 and Day 8. Participants will leave the CPC following completion of all procedures on Day 12.

Participants will return to the CPC for a final visit 7 (±1) days after their final dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Be capable of and willing to comply with study restrictions and procedures
* Female participants must be non-nursing, have a negative pregnancy test result at screening and Day -1, and be surgically sterile for at least 90 days prior to screening or postmenopausal
* Male participants with female partners of child bearing potential must agree to use 2 acceptable forms of birth control for the duration of the study and for 90 days following the last administration of the drug; all male participants must refrain from donating sperm for this same period
* Be considered healthy by the Investigator, based on participant's reported medical history, full physical examination, clinical laboratory tests, 12-lead electrocardiograms (ECG) and vital signs
* Have normal renal function as determined by Investigator
* Have a body mass index (BMI) of 18.0 to 30.0 kg/m^2 inclusive and body weight >50.0 kg at screening
* Have no relevant dietary restrictions
* Be willing to comply with COVID-19 policy

Exclusion Criteria:

* Clinically significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, renal, hepatic, bronchopulmonary, psychiatric, neurologic, immunologic or lipid metabolism disorders, or drug hypersensitivity as determined by the Investigator
* Known or suspected malignancy
* History of pancreatitis or gall stones
* History of unexplained syncope, symptomatic hypotension, or hypoglycemia
* Personal or family history of long QTc syndrome; QTcF >450 ms
* History of chronic diarrhea, malabsorption, unexplained weight loss, food allergies or intolerance
* Gastrointestinal, liver, kidney disease, or other diseases known to interfere with drug absorption, distribution, metabolism, or excretion within 3 months prior to the screening and during the screening period
* Hypersensitivity to dazucorilant or itraconazole or any components of either formulation
* Poor venous access
* Positive blood screen for infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Donated or lost ≥500 mL of blood in the previous 60 days
* Plasma donation within 30 days prior to the 1st dose of study medication
* Taken an investigational drug or participated in a clinical trial within 90 days (or 5 half-lives), whichever is longer, prior to the 1st dose of study medication
* Used prescription or over-the-counter (OTC) medication (other than ≤1 g/day acetaminophen), antacids, vitamins or herbal remedies or supplements, within 2 weeks or 5 half-lives before first study drug administration, whichever is longer
* Used food or drugs that are inducers of CYP3A4/5 and/or P-glycoprotein inducers within 30 days prior to the first dose of study medication
* Consumption of grapefruit, pomelo, or Seville oranges or their juices or jams, from 30 days prior to Day -1
* Hospital admission or major surgery within 6 months prior to screening or a preplanned hospital admission during study participation
* A history of prescription drug abuse or illicit drug use within 12 months prior to screening
* Use of cannabis or cannabidiol (CBD) containing products within 30 days prior to study drug administration on Day 1
* A history of alcohol abuse according to medical history within 2 years prior to screening
* Use of tobacco- or nicotine-containing products or participants unwilling/unable to stop nicotine intake from 6 months prior to screening until the end of the study
* A positive screen for alcohol, drugs of abuse, or cotinine at screening or Day -1
* An unwillingness or inability to comply with food and beverage restrictions during study participation
* Investigational site staff members directly involved in the conduct of the study and their family members; site staff members otherwise supervised by the Investigator or Corcept Therapeutics Incorporated employees directly involved in the conduct of the study
* Any condition or finding that in the Investigator's opinion would put the participant or study conduct at risk if the participant were to participate in the study
* Unable to complete this study for other reasons or the Investigator believes that he or she should be excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2024-05-31 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of dazucorilant | Predose and at serial timepoints up to 96 hours after dazucorilant dosing on Days 1 and 8
Area under the concentration-time curve from time 0 to the last measurable concentration (AUClast) of plasma dazucorilant | Predose and at serial timepoints up to 96 hours after dazucorilant dosing on Days 1 and 8
Area under the concentration-time curve from time 0 extrapolated to infinity (AUCinf) of plasma dazucorilant | Predose and at serial timepoints up to 96 hours after dazucorilant dosing on Days 1 and 8

SECONDARY OUTCOMES:
Number of Participants with 1 or More Adverse Events | Up to Day 18
Number of Participants with 1 or More Clinically Significant Abnormal ECG Result | Up to Day 18
Number of Participants with 1 or More Clinically Significant Abnormal Vital Signs | Up to Day 18
Number of Participants with 1 or More Clinically Significant Abnormal Physical Examination Finding | Up to Day 18
Number of Participants with 1 or More Clinically Significant Abnormal Clinical Laboratory Test Result | Up to Day 18

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Custodio, PhD, Study Director — Corcept Therapeutics
Locations (1):
- Site 01, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No